CLINICAL TRIAL: NCT06182852
Title: An Observational Clinical Study on the Effect of GLP-1 Receptor Agonist on Bone Metabolism in Patients With Diabetes Mellitus
Brief Title: The Effect of GLP-1 Receptor Agonist on Bone Metabolism in Patients With Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20231109-08
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-11

CONDITIONS: Diabete Type 2; Bone Metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- glucagon-like peptide-1receptor agonists: Once a week, hypodermic injection.

SUMMARY:
Through an one-year follow-up, to explore the effect of GLP-1 receptor agonist on bone metabolism in patients with diabetes.

DETAILED DESCRIPTION:
This study is a single-center observational study. After the patients were enrolled according to the standard of admission and exclusion, on the basis of the original scheme, GLP-1 receptor agonists were added and followed up for one year. The indexes of bone metabolism and body fat were measured at several time points (3 months, 6 months, 9 months and 12 months after treatment). Bone mineral density (BMD) was measured at several time points (6 months and 12 months after treatment) to explore the effect of GLP-1 receptor agonists on bone metabolism in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed patients with diabetes
2. HbA1c≥7.5%；
3. Willing to sign a written informed consent form and abide by the research plan

Exclusion Criteria:

1. Any of the following drugs or treatments were used within one month before screening: treated with GLP-1RA, GLP-1 analogues, DPP-4 inhibitors, or any other enterotropic insulin analogue
2. Long-term intravenous, oral and intra-articular administration of corticosteroids within 2 months before screening (more than 7 days in a row)
3. Use of weight control drugs or surgery that can lead to weight instability within the first 2 months of screening, or are currently in the weight loss plan and are not in the maintenance stage
4. History of acute and chronic pancreatitis; history of myeloid C cell carcinoma, MEN (multiple endocrine tumors) 2A or 2B syndrome, or related family history
5. There is a clinically significant abnormal gastric emptying.
6. Screening of any organ system tumors that have been treated or untreated within the previous 5 years
7. Underwent coronary angioplasty, coronary stent implantation and coronary artery bypass surgery within 6 months before selection, resulting in negligent compensatory heart failure (New York Heart Association NYHA classification III and IV), stroke or transient ischemic attack, unstable angina pectoris, myocardial infarction, persistent and clinically significant arrhythmias.
8. Acute metabolic complications occurred within 6 months before screening. （9）Before screening, any laboratory test index meets the following criteria: glutamic pyruvic transaminase > 2.5 times or aspartate oxaloacetic transaminase > 2.5 times; eGFR < 45ml < 45ml hand minmax 1.73m2; fasting triglyceride > 5.64mmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Diagnosed patients with diabetes
  2. HbA1c≥7.5%
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Bone metabolism | 3、6、9、12month
  Changes of bone metabolic indexes before and after treatment
Bone mineral density | 6、12month
  Changes of bone mineral density before and after treatment
HbA1c | 0、3、6、9、12month
  the glycosylated hemoglobin level of patients

SECONDARY OUTCOMES:
Body fat | 3、6、9、12month
  The changes of body fat mass after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing Medical Univesity, Nanjing, Nanjing,, China